CLINICAL TRIAL: NCT01506830
Title: Influence of Operatory Field Isolation Techniques on the Clinical Performance of Class V Restorations
Brief Title: Cervical Restorations Placed Under Two Isolation Methods
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Federal University of Pelotas (Other)
Responsible Party: Principal Investigator, Maximiliano Sergio Cenci, PhD, Coordinator of Clinical Trials, Graduate Program in Dentistry, Federal University of Pelotas
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UFPEL-PPGO0012
Record Dates: First submitted 2011-12-30; First posted 2012-01-10 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Non-carious Cervical Lesions
Keywords: Adhesives.; Composites.; Noncarious cervical lesions.; Clinical performance.; Treatment
MeSH Terms: interventions — Rubber Dams

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Absolute isolation (Active Comparator): Absolute isolation of the operatory field with rubber dam: Moisture control is provided by a rubber dam and a gingival retraction clamp placed in the cervical area of the tooth.
  Interventions: Procedure: Absolute isolation with rubber dam
- Relative isolation (Experimental): Relative isolation of the operatory field with cotton rolls: Moisture control was provided using a labial retractor, cotton rolls and gingival retraction cord placed into the gingival sulcus
  Interventions: Procedure: Relative isolation with cotton rolls

INTERVENTIONS:
Procedure: Relative isolation with cotton rolls — Cotton roll group: Moisture control was provided using a labial retractor, cotton rolls and gingival retraction cord placed into the gingival sulcus
  Arms: Relative isolation
Procedure: Absolute isolation with rubber dam — Rubber dam group: Moisture control was provided by a rubber dam and a gingival retraction clamp placed in the cervical area of the tooth.
  Arms: Absolute isolation

SUMMARY:
During restorative procedures, different isolation methods of the operative field can be used to promote moisture control and retraction of the gingival tissues. The aim of the present clinical trial is to evaluate the effects of two isolation techniques on the clinical performance of Class V restorations, as well on the periodontal conditions of restored sites. Patients presenting at least two noncarious cervical lesions (NCLs) will be enrolled in this study. The NCLs will be randomized into the following groups: (1) isolation performed with rubber dam and gingival retraction clamp and (2) isolation provided with cotton rolls and gingival retraction cord. Both techniques will be used with a saliva suction device. All restorative procedures were performed using a self-etching adhesive system and a nanofilled composite resin according to the manufacturer's instructions. The clinical performance of restorations will be recorded in terms of fracture and retention of restoration, marginal adaptation, marginal staining, postoperative hypersensitivity, and preservation of tooth vitality at 1 week, 6 months, 12, 24 and 72 months after placement. The periodontal condition of restored sites will be evaluated based on the presence of supragingival plaque, gingival marginal bleeding, probing depth, and relative gingival recession.

ELIGIBILITY:
Inclusion Criteria:

* more than one cervical lesion
* lesions whose apical limit located above the gingival margin
* lesions with at least 1 mm of depth
* vital permanent incisors, canines, or premolars

Exclusion Criteria:

* smoking habits
* severe systemic diseases
* active orthodontic treatment
* malocclusion (Angle Class II or Class III)
* less than 20 natural teeth in mouth
* absent of antagonist tooth
* wear facets over more than 50% of the incisal/occlusion surface as a result of tooth attrition
* or restorations in the area to be treated
* full-mouth visible plaque index (VPI) or full-mouth gingival bleeding index (GBI) more than 20%
* probing depth (PD) and clinical attachment loss (CAL) values exceeding 4 mm with bleeding on probing (BOP)
* unwillingness to return for follow-ups or refuse to participate

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-07; Primary Completion 2011-07 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
retention of restorations | up to 72 months
  Retention of restorations is measured by clinical examination, where each placed restoration is checked and scored as present, partially lost or lost at the recalls.
Restorations marginal staining | up to 72 months
  Restorations are checked during recalls regarding the marginal staining and scored as clinically ideal, clinically acceptable; presence of small ditching; presence of extensive marginal ditching and need for repair /replacement.

SECONDARY OUTCOMES:
Periodontal condition of restored sites | 6, 12, 24, 48 and 72 months after restorations' placement
  The periodontal condition of restored sites is evaluated based on the presence of supragingival plaque, gingival marginal bleeding, probing depth, and relative gingival recession.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre S Masotti, PhD, Study Chair — Federal University of Pelotas; Fernanda OB Corrêa, PhD, Principal Investigator — Federal University of Pelotas; Silvia T Fontes, PhD, Principal Investigator — Federal University of Pelotas; Maximiliano S Cenci, PhD, Principal Investigator — Federal University of Pelotas; Patricia S Jardim, PhD, Principal Investigator — Federal University of Pelotas
Locations (1):
- Federal University of Pelotas - School of Dentistry, Pelotas, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Favetti M, Montagner AF, Fontes ST, Martins TM, Masotti AS, Jardim PDS, Correa FOB, Cenci MS, Muniz FWMG. Effects of cervical restorations on the periodontal tissues: 5-year follow-up results of a randomized clinical trial. J Dent. 2021 Mar;106:103571. doi: 10.1016/j.jdent.2020.103571. Epub 2020 Dec 29. PMID 33385534